CLINICAL TRIAL: NCT01990560
Title: Glucocorticoid Receptor Blockade With Mifepristone in Patients With Mild Adrenal Hypercortisolism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Alice C. Levine, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 13-1061
Record Dates: First submitted 2013-11-15; First posted 2013-11-21 (Estimated); Results first posted 2018-03-02 (Actual); Last update posted 2018-03-02 (Actual); Status verified 2018-01

CONDITIONS: Mild Hypercortisolism
Keywords: mild hypercortisolism; Subclinical Cushing's Syndrome; Preclinical Cushing's Syndrome
MeSH Terms: interventions — Mifepristone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mifepristone (Experimental): Mifepristone 300mg tablets taken once daily with dose increase of no more than 300mg once monthly and to a maximum dose of 1200mg daily as indicated by symptom response
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone — All patients in the study will receive daily Mifepristone for 6 months and primary and secondary outcomes will be assessed before and after the 6 month treatment period
  Other Names: Korlym

SUMMARY:
The purpose of this study is to determine whether mifepristone is an effective treatment for hyperglycemia due to mild hypercortisolism.

* To test the hypothesis that GR blockade with mifepristone will decrease the severity of metabolic syndrome features as measured by waist circumference, lipid profile, body mass index, blood pressure and insulin resistance, measured by HOMA-IR score.
* To test the hypothesis that GR blockade with mifepristone will improve QoL, depression and anxiety scores, measured by validated assessments, in patients with mild hypercortisolism.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Incidentally noted adrenal nodule <4 cm with benign imaging characteristics
* Evidence of mild hypercortisolism
* Evidence of diabetes or abnormal glucose tolerance

Exclusion Criteria:

* contraindication to mifepristone
* Indication for unilateral adrenalectomy
* Evidence of other adrenal hormone hypersecretion
* lactating mothers
* women of childbearing age unwilling to use an effective, nonhormonal form of contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice C Levine, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Background] Young WF Jr. Management approaches to adrenal incidentalomas. A view from Rochester, Minnesota. Endocrinol Metab Clin North Am. 2000 Mar;29(1):159-85, x. doi: 10.1016/s0889-8529(05)70122-5. PMID 10732270
- [Background] Mansmann G, Lau J, Balk E, Rothberg M, Miyachi Y, Bornstein SR. The clinically inapparent adrenal mass: update in diagnosis and management. Endocr Rev. 2004 Apr;25(2):309-40. doi: 10.1210/er.2002-0031. PMID 15082524
- [Background] Tauchmanova L, Rossi R, Biondi B, Pulcrano M, Nuzzo V, Palmieri EA, Fazio S, Lombardi G. Patients with subclinical Cushing's syndrome due to adrenal adenoma have increased cardiovascular risk. J Clin Endocrinol Metab. 2002 Nov;87(11):4872-8. doi: 10.1210/jc.2001-011766. PMID 12414841
- [Background] Terzolo M, Pia A, Ali A, Osella G, Reimondo G, Bovio S, Daffara F, Procopio M, Paccotti P, Borretta G, Angeli A. Adrenal incidentaloma: a new cause of the metabolic syndrome? J Clin Endocrinol Metab. 2002 Mar;87(3):998-1003. doi: 10.1210/jcem.87.3.8277. PMID 11889151
- [Background] Garrapa GG, Pantanetti P, Arnaldi G, Mantero F, Faloia E. Body composition and metabolic features in women with adrenal incidentaloma or Cushing's syndrome. J Clin Endocrinol Metab. 2001 Nov;86(11):5301-6. doi: 10.1210/jcem.86.11.8059. PMID 11701696
- [Background] Feelders RA, Hofland LJ. Medical treatment of Cushing's disease. J Clin Endocrinol Metab. 2013 Feb;98(2):425-38. doi: 10.1210/jc.2012-3126. Epub 2013 Jan 23. PMID 23345100
- [Background] Lambert JK, Goldberg L, Fayngold S, Kostadinov J, Post KD, Geer EB. Predictors of mortality and long-term outcomes in treated Cushing's disease: a study of 346 patients. J Clin Endocrinol Metab. 2013 Mar;98(3):1022-30. doi: 10.1210/jc.2012-2893. Epub 2013 Feb 7. PMID 23393167
- [Background] Neary NM, Booker OJ, Abel BS, Matta JR, Muldoon N, Sinaii N, Pettigrew RI, Nieman LK, Gharib AM. Hypercortisolism is associated with increased coronary arterial atherosclerosis: analysis of noninvasive coronary angiography using multidetector computerized tomography. J Clin Endocrinol Metab. 2013 May;98(5):2045-52. doi: 10.1210/jc.2012-3754. Epub 2013 Apr 4. PMID 23559084
- [Background] Debono M, Chadarevian R, Eastell R, Ross RJ, Newell-Price J. Mifepristone reduces insulin resistance in patient volunteers with adrenal incidentalomas that secrete low levels of cortisol: a pilot study. PLoS One. 2013;8(4):e60984. doi: 10.1371/journal.pone.0060984. Epub 2013 Apr 5. PMID 23577182
- [Background] Nieman LK, Biller BM, Findling JW, Newell-Price J, Savage MO, Stewart PM, Montori VM. The diagnosis of Cushing's syndrome: an Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2008 May;93(5):1526-40. doi: 10.1210/jc.2008-0125. Epub 2008 Mar 11. PMID 18334580
- [Background] Flint A, Raben A, Blundell JE, Astrup A. Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies. Int J Obes Relat Metab Disord. 2000 Jan;24(1):38-48. doi: 10.1038/sj.ijo.0801083. PMID 10702749
- [Background] Parker BA, Sturm K, MacIntosh CG, Feinle C, Horowitz M, Chapman IM. Relation between food intake and visual analogue scale ratings of appetite and other sensations in healthy older and young subjects. Eur J Clin Nutr. 2004 Feb;58(2):212-8. doi: 10.1038/sj.ejcn.1601768. PMID 14749739

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mifepristone
Started | 8
Completed | 7
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Mifepristone
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: A1C Level
Description: Change in hyperglycemia assessed by HbA1c, also known as glycated hemoglobin
Time Frame: Baseline, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: percentage of red blood cells
Arm/Group | Mifepristone
Number analyzed (Participants) | 8
percentage of red blood cells
  Baseline | 6.2 (0.58)
  3 months | 6.1375 (0.49)
  6 months | 6.125 (0.72)

2. Primary Outcome: HOMA-IR
Description: Change in hyperglycemia assessed by Homeostatic Model Assessment of Insulin Resistance, HOMA-IR (a validated assessment of insulin resistance). HOMA-IR = fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5.
Time Frame: Baseline and 6 months
Population: one participant on insulin. another participant had data missing at 6 months.
Measure: Mean (Standard Deviation); unit: HOMA-IR score
Arm/Group | Mifepristone
Number analyzed (Participants) | 6
HOMA-IR score
  Baseline | 2.418 (1.64)
  6 months | 1.465 (1.19)

3. Secondary Outcome: Waist Circumference
Description: Change in metabolic syndrome as assessed by waist circumference
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Mifepristone
Number analyzed (Participants) | 8
cm
  Baseline | 103.25 (17.43)
  6 months | 99.3125 (101.25)

4. Secondary Outcome: Body Mass Index (BMI)
Description: Change in metabolic syndrome as assessed by BMI
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Mifepristone
Number analyzed (Participants) | 8
kg/m2
  Baseline | 35.1538 (15.02)
  6 months | 34.5463 (15.84)

5. Secondary Outcome: Fasting Lipid Profile
Description: Change in metabolic syndrome as assessed by fasting lipid profile which includes Low-density lipoproteins ( LDL), High-density lipoproteins (HDL), and Triglycerides (Trigs) levels, and total cholesterol which is the sum of HDL plus LDL and 20% of trigs.
Time Frame: Baseline and 6 months
Population: one participant data missing at 6 month
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Mifepristone
Number analyzed (Participants) | 8
mg/dL
  Total Cholesterol Baseline | 178.63 (31.35)
  Total Cholesterol 6 months: number analyzed (Participants) | 7
  Total Cholesterol 6 months | 171.43 (54.62)
  LDL baseline | 97.88 (22.34)
  LDL 6 months: number analyzed (Participants) | 7
  LDL 6 months | 104.37 (44.69)
  HDL Baseline | 59.13 (19.50)
  HDL 6 months: number analyzed (Participants) | 7
  HDL 6 months | 46.86 (14.26)
  Trigs Baseline | 107.88 (43.90)
  Trigs 6 months: number analyzed (Participants) | 7
  Trigs 6 months | 100.29 (20.21)

6. Secondary Outcome: Weight
Description: Change in metabolic syndrome as assessed by weight
Time Frame: Baseline and 6 months
Population: one participant had data missing at 6 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Mifepristone
Number analyzed (Participants) | 8
kg
  Baseline | 99.57 (38.68)
  6 months: number analyzed (Participants) | 7
  6 months | 97.75 (41.15)

7. Secondary Outcome: CushingQoL
Description: Change in Quality of Life - as assessed by the Cushing's Quality of Life questionnaire (CushingQoL). Patient completed questionnaire, 12 items, each scored on a 5 point score, resulting in a score of 12 (worst) to 60 (best) where higher scores indicate more favorable QOL.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mifepristone
Number analyzed (Participants) | 7
units on a scale
  Baseline | 37.2857 (9.86)
  6 months | 38.7857 (10.20)

8. Secondary Outcome: Nottingham Health Profile (NHP)
Description: Change in Quality of Life as assessed by the Nottingham Health Profile (NHP) which is a patient reported questionnaire to measure a patient's view of their own health status. There are 6 sections (Energy level, Pain, Emotional Reaction, Sleep, Social Isolation, and Physical Abilities. All questions have only yes/no answer options and each section score is weighted so that the possible score range for any section is 0-100. The higher the score, the greater the number and severity of problems.
Time Frame: Baseline and 6 months
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Mifepristone
Number analyzed (Participants) | 7
units on a scale
  Energy Level (EL) Baseline | 32.60 [0 to 38]
  EL 6 months | 45.40 [18 to 72.4]
  Pain (P) Baseline | 24.88 [0 to 25.1]
  P 6 months | 32.08 [0 to 44.5]
  Emotional Reaction (ER) Baseline | 27.03 [0 to 38.7]
  ER 6 months | 35.09 [7.3 to 54.6]
  Sleep (S) Baseline | 24.87 [5.4 to 38.8]
  S 6 months | 31.15 [0 to 46.3]
  Social Isolation (SI) Baseline | 20.09 [0 to 21]
  SI 6 months | 31.15 [0 to 46.29]
  Physical Abilities (PA) Baseline | 23.06 [0 to 48.2]
  PA 6 months | 27.49 [17.6 to 42.2]

9. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: Change in Quality of Life as assessed by the Hospital Anxiety and Depression Scale (HADS). Questionnaire with 7 items for anxiety and 7 items for depression, each item is scored on a 4 point response 0 - 3, with full range from 0 to 42, with higher score indicating more severe anxiety or depression
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mifepristone
Number analyzed (Participants) | 7
units on a scale
  Baseline | 16.2857 (10.90)
  6 months | 11.1667 (8.23)

10. Secondary Outcome: Quality of Life
Description: Change in Quality of Life as assessed by the Beck Depression Inventory. a 21-question multiple choice, self-report inventory that is used for measuring the severity of anxiety. Scoring is from a 0 (not at all) to 3 (severe) with a total score range of 0-63. Higher total scores indicate more severe anxiety symptoms.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mifepristone
Number analyzed (Participants) | 7
units on a scale
  Baseline | 16.1429 (10.32)
  6 months | 11.7143 (11.70)

11. Secondary Outcome: State Trait Anxiety Inventory (STAI)
Description: Change in Quality of Life - as assessed by the State Trait Anxiety Inventory (STAI). The State-Trait Anxiety Inventory both state and trait anxiety separately. Each type of anxiety has its own scale of 20 different questions that are scored and averaged. Total scores range from 20 to 80, with higher scores correlating with greater anxiety.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mifepristone
Number analyzed (Participants) | 7
units on a scale
  Baseline | 25.4286 (17.61)
  6 months | 28.8571 (10.92)

ADVERSE EVENTS:
Arm/Group | Mifepristone
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mifepristone (N=8)
Drug Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes